CLINICAL TRIAL: NCT05625139
Title: Implementation of an Enhanced Rehabilitation Protocol After Liver Transplantation: Feasibility and Analysis of Results
Acronym: IPRA
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7906
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2022-11

CONDITIONS: Liver Transplant Disorder
Keywords: Liver Transplant Disorder; Liver transplantation; ERAS

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Currently, there are no expert recommendations regarding enhanced rehabilitation after liver transplantation. The development of Enhanced Rehabilitation After Surgery (ERAS) protocols in major surgery, particularly cardiothoracic surgery, has motivated some anesthesia teams to extubate liver transplant patients earlier who meet predefined criteria (young patient, absence of comorbidities, absence of intraoperative transfusion) in order to limit the occurrence of complications of mechanical ventilation (pneumopathies, tracheal wound, muscle loss, etc.) On the other hand, improved rehabilitation in this case was often synonymous with early extubation in the operating room. Few studies, on the other hand, relate the implementation of a complete rehabilitation protocol including pre-, intra- and postoperative guidelines.

ELIGIBILITY:
Inclusion criteria:

* Major subject operated at HUS for a liver transplant whose management was scheduled in the Surgical Intensive Care Unit fbetween December 01, 2018 and August 31, 2020
* Subject who does not question, after information, the reuse of his data for the purpose of this research

Exclusion criteria:

* Subject having expressed his opposition to participate in the study
* Liver transplant patient hospitalized in the Medical Intensive Care Unit before or after the surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject operated at HUS for a liver transplant whose management was scheduled in the Surgical Intensive Care Unit fbetween December 01, 2018 and August 31, 2020
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-11-14 (Actual)

PRIMARY OUTCOMES:
Retrospective description of the protocol of improved rehabilitation after liver transplantation, to study the possibility of its implementation in the anesthesia-intensive care department and to analyze the first results | Files analysed retrospectively from December 01, 2018 to August 31, 2020 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie, Réanimation et Médecine péri-Opératoire - CHU de Strasbourg - France, Strasbourg, France